CLINICAL TRIAL: NCT04101240
Title: Impact of Perioperative Anemia and Red Blood Cells Transfusion on Post-operative Complications After Oncological Surgery
Brief Title: Anemia and Red Blood Cells Transfusion in Oncological Surgery
Acronym: IMPACT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: IMPACT (29BRC19.0013)
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Anemia; Surgery; Oncology
Keywords: red blood cells transfusion
MeSH Terms: conditions — Anemia; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Oncologic patients experience anemia and anemia is associated with poor prognosis. Transfusion is associated with adverse events, and equipoise remains on the optimal transfusion strategy in oncologic patients in surgical setting. The primary objective of this study is to determine the impact of anemia and red blood cells (RBC) transfusion on post-operative complications and mortality.

DETAILED DESCRIPTION:
Between 36 and 75% of oncologic patients experience anemia and anemia is associated with poor prognosis. Up to 40% of surgical oncologic patients receive red blood cells (RBC). However, transfusion is associated with adverse events, and equipoise remains on the optimal transfusion strategy in oncologic patients in surgical setting. The primary objective of this study is to determine the impact of anemia and red blood cells (RBC) transfusion on post-operative complications and mortality. This is a retrospective, single center study. All adults admitted to the intensive care unit (ICU) after oncologic surgery within the study period are eligible.

ELIGIBILITY:
Inclusion Criteria:

* Surgery for cancer
* Admission to intensive care

Exclusion Criteria:

* no consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults admitted to the intensive care unit (ICU) after oncologic surgery from January 2017 to December 2018 are eligible. The following types of surgery for cancer or metastasis resection with a high risk of bleeding are eligible: thoracic, abdominal, neurosurgery, gynecologic, urologic, otorhinolaryngology or spinal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-07 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of mortality or any respiratory, cardiac, renal, thromboembolic, infectious and/or hemorrhagic post operative complications | 30 DAYS (hospital discharge)
  mortality or any respiratory, cardiac, renal, thromboembolic, infectious and/or hemorrhagic post operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Cécile AUBRON, PU PH, Principal Investigator — Service de Médecine Intensive Réanimation
Locations (1):
- CHRU de Brest, hôpital de la Cavale Blanche, Brest, France